CLINICAL TRIAL: NCT04507633
Title: The Effect of ROMA Therapy on Improving Cognitive Functions, Depressive Symptoms and Behavioral Problems in the Population With Dementia
Brief Title: ROMA (Reminiscence, Reality Orientation, Music and Art ) Therapy, Cognition, Depression and Behavioral Problems in the Population With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Huang, Hui-Chuan, Associate Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: N202005108
Record Dates: First submitted 2020-07-25; First posted 2020-08-11 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia | interventions — Reproductive Techniques, Assisted

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: independent researchers will perform intervention and data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ROMA therapy (Experimental): ROMA therapy combines four elements including reminiscence, reality orientation, music, and art in the intervention.
  Interventions: Behavioral: ROMA therapy(reminiacence therpy, orientation, music, and art)
- control group (No Intervention): usual care

INTERVENTIONS:
Behavioral: ROMA therapy(reminiacence therpy, orientation, music, and art) — An intervention comprising reminiscence of annual festivals, orientation, and familiar music listening and singing, and animation interaction to improve cognitive functions, depressive symptoms and behaviors problems.
  Arms: ROMA therapy

SUMMARY:
This study aimed to conduct a randomized controlled trial to examine the effectiveness of ROMA therapy( Reminiscence, Reality Orientation, Music, and Art) on improving cognitive function, behavioral and psychological symptoms in population with dementia. The hypotheis of this study is that these patients with dementia receiving ROMA therapy featuring reminiscence, reality orientation, music, and art would improve their cognition, depressive symptoms, and behavioral symptoms.

DETAILED DESCRIPTION:
This study aimed to conduct a randomized controlled trial to examine the effectiveness of ROMA therapy( Reminiscence, Reality Orientation, Music, and Art) on improving cognitive function, behavioral and psychological symptoms in demented population. A total of 60 patients with mild to moderate dementia will be recruited and randomly assigned to two groups: experimental group and control group. The experimental group will undergo ROMA therapy with a 60 minute per week for eight weeks. The control group will receive three times ROMA therapy after completing outcome measurements. Two groups will receive questionnaire interview at pre-test, post-test, and at 4 weeks after intervention. The measurements comprises: Short Portable Mental Status Questionnaire(SPMSQ), Cornell Scale for Depression in Dementia(CSDD),and Neuropsychiatric Inventory-Questionnaire(NPI-Q). By identifying the effectiveness of ROMA therapy, suitable intervention can be suggested for those demented population to improve cognitive function, behavioral and psychological symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Been diagnosed as mild to moderate dementia and CDR score between 0.5~2
2. can communicate in Chinese or Taiwanese
3. without visual or auditory impairment after equipping assist devices

Exclusion Criteria:

1. severe dementia and Clinical Dementia Rating (CDR) score more than 2 points
2. functional dependence
3. incapable of expressing their feelings

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
cognitive functions | cognitive functions at baseline
  Short Portable Mental Status Questionnaire(SPMSQ)
cognitive functions | cognitive functions after the completion of intervention
  Short Portable Mental Status Questionnaire(SPMSQ)
cognitive functions | cognitive functions at 4 weeks after the completion of intervention
  Short Portable Mental Status Questionnaire(SPMSQ)
depressive symptoms | depressive symptoms at baseline
  Cornell Scale for Depression in Dementia(CSDD)
depressive symptoms | depressive symptoms after the completion of intervention
  Cornell Scale for Depression in Dementia(CSDD)
depressive symptoms | depressive symptoms at 4 weeks after the completion of intervention
  Cornell Scale for Depression in Dementia(CSDD)
behavioral problems | behavioral problems at baseline
  Neuropsychiatric Inventory-Questionnaire(NPI-Q)
behavioral problems | behavioral problems after the completion of intervention
  Neuropsychiatric Inventory-Questionnaire(NPI-Q)
behavioral problems | behavioral problems at 4 weeks after the completion of intervention
  Neuropsychiatric Inventory-Questionnaire(NPI-Q)

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Chuan Huang, PhD, Principal Investigator — School of Nursing, Taipei Medical University
Locations (1):
- Yonghe Zhongxing Public Seniors Center, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tz-Han L, Wan-Ru W, I-Hui C, Hui-Chuan H. Reminiscence music intervention on cognitive, depressive, and behavioral symptoms in older adults with dementia. Geriatr Nurs. 2023 Jan-Feb;49:127-132. doi: 10.1016/j.gerinurse.2022.11.014. Epub 2022 Dec 8. PMID 36495795